CLINICAL TRIAL: NCT00286299
Title: Physiological and Psychiatric Effects From Aerobic High Intensity Endurance Training and Maximal Strength Training in Patients Suffering From Schizophrenia: A Controlled Clinical Trial.
Brief Title: Treatment Effects From Aerobic Endurance Training and Maximal Strength Training in Patients Suffering From Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2005.1507
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Cardiovascular Disease
Keywords: Schizophrenia; Cardiovascular disease; Aerobic capacity; Mortality; Exercise
MeSH Terms: conditions — Schizophrenia; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic interval training (AIT) (Experimental): AIT is 4x4 minutes interval training on a treadmill at 85 to 95 % HRpeak interspersed with 3 min of active resting periods at a work load corresponding to 70 % HRpeak between each interval. Patients performed the intervals walking or running with a minimum of 5 % inclination.
  Interventions: Other: Aerobic high-intensity interval training (AIT)
- Computer game training (CG) (Active Comparator): 36 minutes playing supervised computer games, Tetris, Xbox
  Interventions: Other: Computer game training (CG)
- Maximal strength training (MST) (Experimental): MST is performed in a leg press machine. The weight is lowered in a controlled manner in the eccentric phase until the patient reached 90 degrees in the knee joint. Then the patients has a short stop (~0.5 second) before the weight is moved as rapidly as possible to complete extension. The training volume is 4 sets of 4RM (i.e. 85-90 % 1RM). The training load is increased with 2.5-5 kg each time patients managed to perform 4 sets with the determined load or each training session.
  Interventions: Other: Maximal strength training

INTERVENTIONS:
Other: Aerobic high-intensity interval training (AIT) — The AIT group trains 4x4 minute interval training on a treadmill at 85-95 % HRpeak interspersed with 3 minutes of active resting periods at a work load corresponding to 70% HRpeak between each interval. All training sessions are monitored and start with a 6 minute warm-up and end with a 5 minute cool-down period at a work load corresponding to 70% HRpeak. Intervals are performed walking or running on a treadmill with a minimum of 5% inclination, 3 times per week for 8 weeks.
  Other Names: 4x4 interval
  Arms: Aerobic interval training (AIT)
Other: Computer game training (CG) — The CG spend the same amount of time (36 minutes), training to improve their ability in the computer game, Tetris. Tetris is a game where small shapes called Tetraminoes fall from the top of the Playfield to the bottom. Players must rotate the Tetraminoes as they fall and fit them together to complete lines. When the player fills an entire line with blocks, that line is removed from the screen. If the player cannot complete lines, the blocks will eventually rise past the top of the screen, and the game ends.
  Other Names: Tetris THQ Inc., Xbox, Microsoft
  Arms: Computer game training (CG)
Other: Maximal strength training — Training starts with a 10 minute warm-up on the treadmill. Maximal strength training is then performed in an inclined leg press machine. The subject lifts 4 maximal repetitions that are repeated 4 times after a 2 minute rest period. Subjects are instructed to lift the weight with an intention of maximal mobilization of force. Training load is increased each time the subject manage to perform 4x4 maximal repetitions. Training is carried out 3 times per week in 8 weeks.
  Other Names: Leg press machine (Technogym); Olympic weights (Eleiko)
  Arms: Maximal strength training (MST)

SUMMARY:
This study investigates treatment effects from aerobic endurance training, maximal strength training and computer game on aerobic capacity, work efficiency and psychiatric symptoms in patients suffering from schizophrenia. The study is a controlled trial. The aim is to describe the population in respect to aerobic capacity and muscular strength. Low aerobic capacity and muscular strength are important risk factors for cardiovascular disease (CVD). The study also aim to evaluate physical and psychiatric effects from physical training. Effects from participation in physical training or computer game on symptoms, depression and quality of life will be investigated. Data will be collected between October 2005 and August 2007.

ELIGIBILITY:
Inclusion criteria: schizophrenia, schizotypal and delusional disorders (F20-F29) according to the international statistical classification of diseases and related health problems, 10th revision (ICD-10) prepared by the World Health Organization. Patients must have stable antipsychotic medication for six weeks prior to participation.

Exclusion criteria: coronary artery disease, chronic obstructive pulmonary disease, not being able to perform physical treadmill testing and exercise, and less than 80% compliance to the training sessions. All subjects go through a physical health examination at inclusion.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
peak aerobic capacity (VO2peak) | Pre- and Posttest

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Pre- and Posttest
Calgary Depression Scale for Schizophrenia (CDSS) | Pre- and Posttest
The 36-item short form (SF-36) | Pre- and Posttest
60 Watt walking efficiency, Net efficiency | Pre- and Posttest
Maximal strength, measured as one repetition maximum (1RM) in a incline leg press machine (Technogym) | Pre- and Post test
Fasting blood samples, systolic and diastolic blood pressure. | Pre- and posttest

CONTACTS AND LOCATIONS:
Overall Officials: Geir Nilsberg, M.D., Study Chair — Norwegian University og Science and Technology; Jørn Heggelund, M.Sc., Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, Department of Psychiatry, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Heggelund J, Nilsberg GE, Hoff J, Morken G, Helgerud J. Effects of high aerobic intensity training in patients with schizophrenia: a controlled trial. Nord J Psychiatry. 2011 Sep;65(4):269-75. doi: 10.3109/08039488.2011.560278. Epub 2011 Feb 18. PMID 21332297